CLINICAL TRIAL: NCT03839472
Title: Continuous Bladder Irrigation Following Transurethral Resection of Bladder Tumors
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Revision to improve cell recovery
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE12818
Record Dates: First submitted 2019-02-08; First posted 2019-02-15 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Non-muscle Invasive Bladder Cancer (NMIBC); Bladder Tumor (TURBT)
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms; Urinary Bladder Neoplasms

STUDY DESIGN:
Intervention Model Description: Single arm where each patient will act as his/her own internal control (cell count before and after CBI).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Continuous Bladder Irrigation (CBI) (Experimental): Each subject will have a TURBT procedure performed per standard of care procedure, which will be followed by the study intervention - Continuous Bladder Irrigation (CBI) for up to two hours after procedure.
  Six samples of discarded bladder irrigation will be collected from each participant (N=20) immediately after TURBT and after the completion of each liter of normal saline 0.9% irrigation (1 to 5 L) for a total of 120 samples.
  Interventions: Procedure: CBI

INTERVENTIONS:
Procedure: CBI — CBI with 5 liters normal saline in 1 liter increments up to 2 hours after TURBT procedure.

SUMMARY:
The purpose of this pilot study is to determine if washing out the bladder with large volumes of saline after surgical removal of bladder tumors helps to decrease the number of loose cells floating within the bladder after surgery. Anticipated decrease in tumor recurrence and/or progression rates will be measured.

DETAILED DESCRIPTION:
Bladder tumor recurrence after resection of non-muscle invasive bladder cancer (NMIBC) occurs in 50-70% of patients despite the use of adjuvant anticancer therapy after surgery. This is a single-arm, non-randomized pilot study looking to determine whether post-Transurethral Resection of Bladder Tumor (TURBT) cells counts differ significantly between continuous washout of the bladder (CBI) with normal saline compared to pre-CBI wash out. Anticipated decrease in tumor recurrence and/or progression rates will also be measured, and each participant will act as their own internal control.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18 years and older diagnosed with a bladder mass on cystoscopy or imaging study
* Primary bladder tumor occurrence

Exclusion Criteria:

* Patients with unresectable bladder tumors, as determined at the time of diagnosis or TURBT , or imaging concerning of T2 or higher disease
* Patients with bladder perforation at the time of TURBT, which is a contraindication to CBI
* Patients from vulnerable populations, including but not limited to impaired subjects, pregnant women, prisoners, family members of the study team
* Any previous history of bladder tumor resection or intravesical chemotherapy/immunotherapy
* History of previous pelvic radiation
* Bladder tumor volume > 5 cm, involvement of prostatic urethra, or any evidence of hydronephrosis on imaging

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Change in mean cells count before versus after liter 1 of CBI | Immediately after CBI procedure.
  The mean cell count obtained before CBI will be compared to the mean cell counts obtained after each liter (5L total) of CBI.
Change in mean cells count before versus after liter 2 of CBI | Immediately after CBI procedure.
  The mean cell count obtained before CBI will be compared to the mean cell counts obtained after each liter (5L total) of CBI.
Change in mean cells count before versus after liter 3 of CBI | Immediately after CBI procedure.
  The mean cell count obtained before CBI will be compared to the mean cell counts obtained after each liter (5L total) of CBI.
Change in mean cells count before versus after liter 4 of CBI | Immediately after CBI procedure.
  The mean cell count obtained before CBI will be compared to the mean cell counts obtained after each liter (5L total) of CBI.
Change in mean cells count before versus after liter 5 of CBI | Immediately after CBI procedure.
  The mean cell count obtained before CBI will be compared to the mean cell counts obtained after each liter (5L total) of CBI.

SECONDARY OUTCOMES:
Recurrence rate of patients who underwent CBI post TURBT. | 2 years after end of treatment
  Participants are followed for additional 2 years during which time, they will receive standard of care. Data collected during their 2-year follow up includes monitoring for recurrence and progression rates.
  Recurrence is defined as the identification of a recurrent tumor of same grade and or stage or lower
Progression rate of patients who underwent CBI post TURBT. | 2 years after end of treatment
  Participants are followed for additional 2 years during which time, they will receive standard of care. Data collected during their 2-year follow up includes monitoring for recurrence and progression rates.
  Progression is defined as a recurrent tumor of higher grade and or stage

CONTACTS AND LOCATIONS:
Overall Officials: Lee Ponsky, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the published article, after deidentification (text, tables, figures).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication
Access Criteria: To be shared with investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose. For individual participant data meta-analysis.